CLINICAL TRIAL: NCT06243809
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Linagliptin 5 mg Film-coated Tablets (LINIPTIN) and Reference Product (Trajenta®) in Healthy Thai Volunteers Under Fasting Conditions
Brief Title: The Bioequivalence Study of Linagliptin 5 mg Film-coated Tablet in Healthy Thai Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BE23-034
Record Dates: First submitted 2024-01-18; First posted 2024-02-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteer
Keywords: Linagliptin
MeSH Terms: interventions — Linagliptin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linagliptin 5 mg, Then Trajenta 5 mg (Experimental): Participants first received Linagliptin 5 mg tablet 1 tablet (Test product) in a fasting state. After a washout period of 1 week, they then received Trajecta 5 mg tablet (Reference product) in a fasting state.
  Interventions: Drug: Linagliptin 5 mg Oral Tablet; Drug: Trajenta 5 MG Oral Tablet
- Trajenta 5 mg, Then Linagliptin 5 mg (Active Comparator): Participants first received Trajenta 5 mg tablet 1 tablet (Reference product) in a fasting state. After a washout period of 1 week, they then recieved Linagliptin 5 mg tablet (Test product) in a fasting state
  Interventions: Drug: Linagliptin 5 mg Oral Tablet; Drug: Trajenta 5 MG Oral Tablet

INTERVENTIONS:
Drug: Linagliptin 5 mg Oral Tablet — Linagliptin 5 mg Oral Tablet
  Other Names: Linagliptin
Drug: Trajenta 5 MG Oral Tablet — Linagliptin 5 mg Oral Tablet (Trajenta )
  Other Names: Linagliptin

SUMMARY:
A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Linagliptin 5 mg Film-coated Tablet (LINIPTIN) and Reference Product (Trajenta®) in Healthy Thai Volunteers under Fasting Conditions

DETAILED DESCRIPTION:
The primary objective of this bioequivalence study is to assess and compare the rate and extent of absorption of a test formulation against a reference formulation, with an additional focus on evaluating the safety profiles of both formulations. This study aims to provide critical insights into the bioequivalence of the two formulations, shedding light on their pharmacokinetic parameters and overall safety in the context of therapeutic efficacy.

Study Design:

A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Linagliptin 5 mg Film-coated Tablet (LINIPTIN) and Reference Product (Trajenta®) in Healthy Thai Volunteers under Fasting Conditions. The crossover design minimizes the impact of inter-individual variability, allowing for a more accurate assessment of the formulations' performance.

Participant Selection:

A total of 48 healthy Thai volunteers will be recruited to participate in the study. The inclusion criteria involve individuals who meet specific health standards and are willing to comply with the study requirements. The emphasis on recruiting healthy volunteers aims to establish a baseline for comparison, ensuring that any observed differences in absorption and safety can be attributed to the formulations under investigation.

Study Conditions:

The study will be conducted under fasting conditions to isolate the impact of the formulations on absorption without interference from food-related variables. Fasting conditions provide a controlled environment to evaluate the formulations' performance and allow for a more accurate determination of bioequivalence.

ELIGIBILITY:
Inclusion Criteria

1. Healthy Thai male subjects between the ages of 18 to 55 years
2. Body mass index between 18.5 to 30.0 kg/m2
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study.
4. Non-pregnant woman (negative pregnancy test) and not currently breast feeding
5. Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 14 days after the end of study in Period 2. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:

   * Postmenopausal for at least 1 year or
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy orhysterectomy) at least 6 months
6. Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 14 days after the end of study in Period 2.
7. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria

1. History of allergic reaction or hypersensitivity to linagliptin or to any of the excipients
2. History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hypo-/hyperthyroid, diabetes), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hyper-/hypotension), psychiatric, neurologic (e.g. seizures), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness
3. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19
4. History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period
5. History or evidence of type 1 diabetes mellitus, diabetic ketoacidosis
6. History or evidence of acute pancreatitis
7. History or evidence of severe infection or severe accident within 14 days prior to check-in in each period
8. History or evidence of severe joint pain
9. History or evidence of bullous pemphigoid
10. History of problems with swallowing tablet or capsule
11. History of sensitivity to heparin or heparin-induced thrombocytopenia
12. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy
13. History of diarrhea, dehydration or vomiting within 24 hours prior to check-in in each period
14. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine)
15. 12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG will be repeated two more times and the average of the three QTc or QRS values will be used to determine the subject's eligibility.
16. Investigation with blood sample shows positive test for HBsAg.
17. Investigation with blood sample shows fasting blood glucose level less than 70 mg/dl or more than 99 mg/dl at screening.
18. Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test
19. Have eGFR (CKD-EPI) < 50 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment.
20. History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study
21. History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.)
22. History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result. In case of alcohol breath test result represents the alcohol concentration range of 1 - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
23. History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study
24. Consume or drink juice of grapefruit or orange or pomelo or its supplement/containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study
25. Use of prescription or nonprescription drugs (e.g. paracetamol, sulfonylureas, insulin, carbamazepine, phenobarbital, phenytoin, ritonavir, rifampicin), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study
26. Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study
27. Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment
28. Subjects with poor venous access or intolerant to venipuncture
29. Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study
30. Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team
31. Subjects who are employees of International Bio Service Co., Ltd., or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-24 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Plasma Area Under the Curve (AUC(0 to 72hr)) for Linagliptin | Through 72 Hours Post Dose
  Plasma Area Under the Curve of Linagliptin
Peak Plasma Concentration (Cmax) of Linagliptin | 72 Hours Post Dose
  Peak Plasma Concentration (Cmax) of Linagliptin

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No